CLINICAL TRIAL: NCT00317434
Title: A Phase I Trial of Lapatinib in Combination With Carboplatin in Patients With Platinum Sensitive Recurrent Epithelial Ovarian Cancer
Brief Title: Maximum Tolerated Dose of Lapatinib When Given With Carboplatin for Recurrent Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to unacceptable non-dose limiting toxicities, excessive treatment delays and limited clinical responses.
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Ronald D. Alvarez, M.D. / Director, Professor - Gynecologic Oncology, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB 0538 - F051025014; 104239
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Lapatinib

INTERVENTIONS:
Drug: lapatinib

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of Lapatinib with Carboplatin AUC 6 in patients with platinum sensitive recurrent ovarian or primary peritoneal carcinoma and to determine the nature and degree of toxicity of Lapatinib in combination with carboplatin AUC 6 in this cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of epithelial ovarian or primary peritoneal cancer
* Measurable disease or evaluable disease with CA125 >100
* One prior treatment with taxane/platinum based chemotherapy, but patients with recurrent ovarian cancer not receiving platinum-based chemotherapy at time of initial diagnosis will be allowed
* Recurrence after treatment free interval of at least 6 mos from completion of primary chemotherapy
* 19 years of age or older
* Life expectancy of greater than 12 weeks
* Performance status of 0, 1 or 2 (based on GOG Performance Status)
* Normal bone marrow, renal and hepatic function based upon lab tests
* Cardiac ejection fraction within institutional normal range
* Ability to swallow and retain oral medication
* Ability to understand a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering study
* Epithelial ovarian tumors of low malignant potential, stromal or germ cell origin
* Non-measurable or non-evaluable disease
* Archived tumor tissue not available for assay
* Patients may not be receiving any other investigational agents or concurrent anticancer therapy, or herbal (alternative) medicines
* Patients with known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent.
* Uncontrolled inter-current illness
* Patients who are pregnant
* HIV-positive patients receiving combination anti-retroviral therapy
* Patients with GI tract disease resulting in an inability to take oral medication

Ages: 19 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-11; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
MTD of Lapatinib measured in cohorts of 3-6 patients each

SECONDARY OUTCOMES:
Clinical response rate defined by RECIST and CA125 values
EGRF, ErbB-2, PTEN and K-ras expression in tissue samples
Correlate serum levels of Lapatinib with AE's & efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D. Alvarez, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Indiana University School of Medicine, Indianapolis, Indiana

REFERENCES:
- [Result] Kimball KJ, Numnum TM, Kirby TO, Zamboni WC, Estes JM, Barnes MN, Matei DE, Koch KM, Alvarez RD. A phase I study of lapatinib in combination with carboplatin in women with platinum sensitive recurrent ovarian carcinoma. Gynecol Oncol. 2008 Oct;111(1):95-101. doi: 10.1016/j.ygyno.2008.07.001. Epub 2008 Aug 8. PMID 18692224